CLINICAL TRIAL: NCT05464264
Title: Deciphering Metacognition and Treatment Response in Depression With a Novel Digital Paradigm
Brief Title: Auditory MMN EEG in TRD in Response to Ketamine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Centre for Addiction and Mental Health (Other); Toronto Metropolitan University (Other)
Responsible Party: Sponsor
Other Study IDs: 22-084
Record Dates: First submitted 2022-06-24; First posted 2022-07-19 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Treatment-resistant Depression (TRD)
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Ketamine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ketamine — Participants suffering from TRD will receive their ketamine treatment intravenously twice weekly for two weeks (4 treatments in total). A dose of 0.5 mg/kg is infused over 40 minutes, with dose adjustments made at the psychiatrist's discretion.

SUMMARY:
To develop and test a neurocomputational model of ketamine treatment response predictions in TRD.

DETAILED DESCRIPTION:
The investigators propose applying a previously validated computational model of the MMN and the ensuing effects of NMDAR antagonism to predict treatment response following ketamine infusions in TRD patients and distinguish ketamine's antisuicidal effects from those related to mood improvements. The study has two subgoals: first, the computational mechanisms underlying MMN reductions that predict ketamine treatment response in TRD patients will be examined. Second, the computational mechanisms will be linked to their underlying neural causes using neural circuit models. Beyond understanding ketamine's short- and long-term mechanisms of action in TRD, the parameters obtained from fitting these models to noninvasive EEG recordings may facilitate single-patient treatment predictions. If successful, this approach may provide clinically useful prognostic statements in individual patients.

ELIGIBILITY:
Inclusion Criteria:

1.18 to 65 years of age 2. Meeting Diagnostic and Statistical Manual for Mental Disorders (DSM-5) criteria for MDD and in a Major Depressive Episode and ≥10 on the Montgomery-Asberg Depression Rating Scale (MADRS).

3. Competent to consent-based on their ability to provide a spontaneous narrative description of the key elements of the study.

4. Failure of at least two trials of antidepressant therapy during the current episode (treatment-resistant depression) and receiving ketamine treatment clinically as administered by their clinician 5. Staying on stable dosages of any concomitant psychotropic medications.

Exclusion Criteria:

1. History of bipolar disorder or psychosis
2. Current substance use or history of substance use during the past year (excluding nicotine and caffeine use disorder)
3. Concomitant major and unstable medical or neurologic illness or a history of seizures.
4. Non-English-speaking individuals.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient participants diagnosed as suffering from a Treatment-Resistant Depression (TRD) that meet the criteria from Diagnosis and Statistical Manual for Mental Disorders (DSM-5), will be eligible to participate in this data collection study. Participants who have agreed to receive ketamine treatments as part of the Interventional Psychiatry Clinical Program at St. Michael's Hospital will be approached and recruited.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Clinical remission | 4 weeks following the baseline visit
  Remission, defined as MADRS <10, and suicide risk reduction is defined as a ≥ 50% reduction in the suicidal ideation item of the MADRS scale from baseline

SECONDARY OUTCOMES:
Modelling | 2 weeks following the baseline visit
  Modelling the underlying cognitive and behavioural mechanisms to their neural causes from the effect of ketamine on TRD patients

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martin J, Gholamali Nezhad F, Rueda A, Lee GH, Charlton CE, Soltanzadeh M, Ladha KS, Krishnan S, Diaconescu AO, Bhat V. Predicting treatment response to ketamine in treatment-resistant depression using auditory mismatch negativity: Study protocol. PLoS One. 2024 Aug 8;19(8):e0308413. doi: 10.1371/journal.pone.0308413. eCollection 2024. PMID 39116153